CLINICAL TRIAL: NCT03603327
Title: Efficacy and Safety of Response Guided Treatment With Direct Acting Anti-Viral Medications for Chronic HCV Infection - A Pilot Study
Brief Title: Response Guided Treatment With Direct Acting Anti-Viral Medications for Chronic HCV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Collaborators: Loyola University, Harel Dahari, PhD, mathematical modeling support (Unknown)
Responsible Party: Principal Investigator, Ohad Etzion, Head of Gastroantrology, Soroka University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0285-17-SOR
Record Dates: First submitted 2018-06-13; First posted 2018-07-27 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Other): All subjects will receive a standard of care treatment- Direct acting anti-viral agents Drugs
  Interventions: Drug: Direct acting anti-viral agents

INTERVENTIONS:
Drug: Direct acting anti-viral agents — Standard of care for Hepatitis C treatment
  Other Names: Treatment

SUMMARY:
To evaluate the efficacy and safety of direct acting anti-viral agents (DAA) therapy in chronically infected Hepatitis C Virus (HCV) patients using an individualized response guided therapy (RGT) model.

DETAILED DESCRIPTION:
Treatment of HCV infection is directed at achieving sustained virological response (SVR), defined as the continued absence of detectable HCV RNA for 12 or more weeks after completion of therapy Given the limited resources available for the costly DAA treatment, implementation of a response-guided treatment (RGT) model to individualize length of DAA therapy in a prospective setting could result in substantial cost saving on HCV drug expenditure in addition to improving patients' compliance to treatment. Furthermore, if adopted at a larger scale, incorporation of such model into clinical practice may enable expansion of access to DAA therapy for patients who are currently not included in the various treatment programs, especially in resource-limited countries.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Clalit insured patients
3. Female and male over the age of 18
4. Capacity to provide written informed consent
5. HCV RNA Viral Load (VL) larger than 105 IU/mL at screening and on at least one other occasion 6 months or more prior to the most recent HCV RNA test result.
6. HCV genotypes 1a, 1b, 2, 3 or 4
7. Liver fibrosis stage 0-4 as determined by one of the following methods performed within 2 years prior to the screening visit:

   1. Fibrotest
   2. Transient elastography
   3. Liver biopsy using the METAVIR scoring system.
8. Patients must have the following laboratory parameters within 3 months of screening

   1. ALT and AST ≤ x10 the upper limit of normal (ULN)
   2. Direct bilirubin ≤ 1.5 the ULN
   3. Platelet count ≥70,000
   4. Hemoglobin ≥10 mg/dL
   5. Albumin ≥3 mg/dL
   6. INR ≤ 1.5 x ULN
   7. eGFR ≥ 60 mL/min as calculated by the Cockroft-Gault equation.
9. Abdominal ultrasound, C.T or MRI scan showing no evidence of a focal lesion suspicious of hepatocellular carcinoma within 6 months of enrollment.
10. A female patient will be eligible to enter the study if it is confirmed that she is:

    1. Not pregnant or nursing
    2. Of non-childbearing potential (following hysterectomy, bilateral oophorectomy or post-menopausal)
    3. Women of childbearing potential- must have a negative urine pregnancy test at baseline and willing to use an accepted mechanical, medical or surgical birth control method from the day of screening until 90 days from the last dose of study drug.
11. All male participants in the study must agree to consistently and correctly use a condom, while their female partner agrees to use one of the above-mentioned birth control methods from the day of screening until 90 days after the last dose of study drug.
12. Patient must be able to comply with the dosing instructions for the study drug administration and able to complete the study schedule of assessments including all required post-treatment visits.

Exclusion Criteria:

1. Clinical, serologic or histopathological evidence supporting the presence of chronic liver disease other than HCV (Including but not limited to: HBV, HDV or HIV coinfection, non-alcoholic steatohepatitis, alcoholic liver disease, Wilson's disease, A1AT deficiency and Celiac disease). Workup performed within 6 months of recruitment will be considered sufficient to exclude the above-mentioned conditions (except for A1AT deficiency and Wilson's disease for which exclusion at any time point qualifies).
2. Current or past history of any of the following:

   1. Clinically significant illness (other than HCV) or any other medical disorder that may interfere with patient's assessment, treatment or compliance with the protocol. Examples include congestive heart disease with moderate to severe left ventricular function and chronic obstructive pulmonary disease requiring chronic corticosteroid therapy.
   2. Clinical evidence of decompensated liver disease (e.g. ascites, bleeding esophageal varices, spontaneous bacterial peritonitis, encephalopathy or hepatorenal syndrome.)
   3. Child Pugh score higher than 6
   4. Gastrointestinal disorder or post-operative condition that may interfere with the absorption of the study drug.
   5. Solid organ transplantation
   6. Malignancy within 5 years prior to screening with the exception of specific cancers that are entirely cured by surgical resection (basal cell skin cancer etc.) Patients under the evaluation for possible malignancy are not eligible.
3. Any prior treatment with a DAA (protease inhibitors, NS5A inhibitors, NS5B polymerase inhibitors/non-nucleoside polymerase inhibitors)
4. Use of anti-viral medications within 30 days of screening.
5. Chronic use of systemically administered immunosuppressive/immune- modulating medications
6. Clinically relevant substance abuse within 6 months of enrollment. Patient with prior history of drug addiction who are currently maintained on a stable dose of opiate substitutes (naloxone) will be allowed to participate in the study if they can provide documentation of repeated negative toxicology screens from the 6 months prior to screening.
7. Participating in clinical trial 30 days before screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of sustained virological response (SVR) | at 12 weeks after the end of treatment in all patients who received at least 4 weeks of therapy with any of the 5 optional drug regimens.
  Sustained virological response (SVR), defined as an HCV RNA level of less than 10 IU/mL and measured by the Cepheid GeneXpert essay.
The percentage of patients in whom duration of treatment with DAA can be shortened to less than 12 weeks. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ohad Etzion, MD, Principal Investigator — Soroka UMC
Locations (2):
- Israel (2):
  - Soroka UMC, Beersheba
  - Rabin Medical Center, Petah Tikva

REFERENCES:
- [Derived] Etzion O, Dahari H, Yardeni D, Issachar A, Nevo-Shor A, Cohen-Naftaly M, Ashur Y, Uprichard SL, Arbib OS, Munteanu D, Braun M, Cotler SJ, Abufreha N, Keren-Naus A, Shemer-Avni Y, Mor O, Murad J, Novack V, Shlomai A. Response guided therapy for reducing duration of direct acting antivirals in chronic hepatitis C infected patients: a Pilot study. Sci Rep. 2020 Oct 20;10(1):17820. doi: 10.1038/s41598-020-74568-x. PMID 33082372